CLINICAL TRIAL: NCT06263192
Title: Pregnancy Prediction in Non-sterile Patients After 4 Intrauterine Inseminations With Donor Using Anti-Müllerian Hormone
Brief Title: Pregnancy Prediction Using Anti-Müllerian Hormone in Intrauterine Insemination Cycles
Status: Completed | Type: Observational
Sponsor: Jose Antonio Moreno (Other)
Collaborators: Universitat Autonoma de Barcelona (Other)
Responsible Party: Sponsor-Investigator, Jose Antonio Moreno, Principal Investigator, Clinica de la Mujer Medicina Reproductiva, Chile
Organization: Clinica de la Mujer Medicina Reproductiva, Chile (Other)
Other Study IDs: AMH-IUI
Record Dates: First submitted 2023-05-11; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Infertility, Female; Anti-Mullerian Hormone Deficiency
Keywords: anti-mullerian hormone; infertility; intrauterine insemination; sperm donation; cumulative pregnancy rates
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AMH < 1.1 ng/ml
  Interventions: Procedure: Intrauterine insemination
- AMH > 1.1 ng/ml
  Interventions: Procedure: Intrauterine insemination

INTERVENTIONS:
Procedure: Intrauterine insemination — Intrauterine insemination with sperm donors

SUMMARY:
The goal of this study is to compare the cumulative pregnancy rates after 4 artificial inseminations with donor (IAD) in non-sterile women with plasma AMH levels > and < 1.1 ng/mL.

ELIGIBILITY:
Inclusion Criteria:

* IUI cycles with sperm donors either due to severe oligoasthenoteratozoospermia in the partner (defined as a motile sperm count (MSC) < 5 million in the ejaculate) or for social reasons, with up to 4 attempts accounted for.

Exclusion Criteria:

* BMI >30
* Infertility due to bilateral tubal factor
* Endometriosis grade II-IV.

Ages: 25 Years to 39 Years | Sex: Female
Age Groups: Adult
Study Population: The study includes all patients between 25 and 39 years of age who have undergone IUI cycles with sperm donors
Sampling Method: Probability Sample
Enrollment: 342 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Cummulative pregnancy rate | 36 months
  Pregnancy rate after 4 cycles of IUI

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Angel Checa, Study Director — Fertty International
Locations (1):
- Fertty International, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gayete-Lafuente S, Moreno-Sepulveda J, Sanchez-Alvarez J, Prat M, Robles A, Espinos JJ, Checa MA. Anti-Mullerian hormone does not predict cumulative pregnancy rate in non-infertile women following four IUI cycles with donor sperm. J Assist Reprod Genet. 2024 Sep;41(9):2319-2326. doi: 10.1007/s10815-024-03188-5. Epub 2024 Jul 10. PMID 38987421